CLINICAL TRIAL: NCT06718712
Title: Effects of Resistance Exercise Volume on the Variability of the Hypertrophic Response in Elderly
Brief Title: Resistance Exercise Volume and Hypertrophic Response Variability in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Hamilton Augusto Roschel da Silva, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 62590416.0.0000.5391
Record Dates: First submitted 2024-12-01; First posted 2024-12-05 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Aging; Muscle Hypertrophy
Keywords: aging; muscle mass; muscle strength; resistance exercise; sets

STUDY DESIGN:
Intervention Model Description: Lower body unilateral design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single set (Experimental): One set of unilateral knee-extension exercise of 8-15 RM with a 60-90 s interval.
  Interventions: Other: Lower body resistance training
- Four sets (Experimental): Four sets of unilateral knee-extension exercise of 8-15 RM with a 60-90 s interval between sets.
  Interventions: Other: Lower body resistance training

INTERVENTIONS:
Other: Lower body resistance training — The RT protocol was performed using a unilateral knee-extension machine. To reduce potential sources of bias to exercise order, subjects alternated the starting leg for each training session.

SUMMARY:
The study aimed to investigate the effects of resistance training volume manipulation on whole muscle hypertrophy among non-responders and responders to a low resistance training dose (single-set).

DETAILED DESCRIPTION:
The magnitude of muscle hypertrophy in response to resistance training (RT) is highly variable between individuals (response heterogeneity). Manipulations in RT variables may modulate RT-related response heterogeneity; yet, this remains to be determined.

ELIGIBILITY:
Inclusion Criteria:

* 60 years and older
* not engaged in regular resistance and/or aerobic training for at least six months before the intervention

Exclusion Criteria:

* diagnosed type I diabetes mellitus
* arrhythmia
* noncontrolled hypertension
* any major orthopedic musculoskeletal condition
* use of any dietary supplement or drug with potential anabolic effects

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Quadriceps muscle cross-sectional area | 10 weeks
  Quadriceps muscle CSA was obtained through magnetic resonance imaging.

SECONDARY OUTCOMES:
Maximum dynamic strength | 10 weeks
  Unilateral quadriceps 1-RM of both legs were assessed on a knee-extension machine

OTHER OUTCOMES:
Dietary assessment | Before intervention
  Dietary assemment using the USDA Automated Multiple-Pass Method
Mass spectrometry | 10 weeks
  Mass spectrometry metabolomics
Skeletal muscle RNA-sequencing | 10 weeks
  RNA sequencing using an Illumina NovaSeq Platform with a standard paired-end 150 bp (PE150) dual indexing protocol
Muscle protein measures | 10 weeks
  Upstream binding factor (UBF) muscle protein was quantified by Simple Western capillary immunoassay.
Muscle protein measures | 10 weeks
  v-Myc Avian Myelocytomatosis Viral Oncogene Homolog (c-Myc) muscle protein was quantified by Simple Western capillary immunoassay.
Muscle protein measures | 10 weeks
  Frizzled class receptor 1 (Frizzled-1) muscle protein was quantified by Simple Western capillary immunoassay.
Muscle protein measures | 10 weeks
  ribosomal protein L3 (rpL3) muscle protein was quantified by Simple Western capillary immunoassay.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No